CLINICAL TRIAL: NCT06441591
Title: The Effect of Vinpocetine on the Clinical Outcome of Patients With Diabetic Nephropathy
Brief Title: Clinical Outcome of Vinpocetine in Diabetic Nephropathy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Salma Hesham Bahram, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 238
Record Dates: First submitted 2024-05-27; First posted 2024-06-04 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Kidney Disease; Diabetic Nephropathies
Keywords: Vinpocetine; Diabetic nephropathy; diabetic kidney disease; UACR; ICAM
MeSH Terms: conditions — Diabetic Nephropathies | interventions — vinpocetine; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vinpocetine + Standard Therapy (Experimental): Vinpocetine capsules, 30 mg, twice daily, with meals for 3 months
  Interventions: Drug: Vinpocetine; Drug: Standard Therapy
- Placebo + Standard Therapy (Placebo Comparator): Placebo, twice daily, with meals for 3 months
  Interventions: Drug: Standard Therapy; Other: Placebo

INTERVENTIONS:
Drug: Vinpocetine — Vinca derivative of apovincamine, phosphodiestrase 1 inhibitor, sodium-gated voltage channel
  Arms: Vinpocetine + Standard Therapy
Drug: Standard Therapy — Anti-hypertensive and anti-diabetic medications according to the the institution's protocol
Other: Placebo — Starch-filled capsules, matching those of the intervention
  Arms: Placebo + Standard Therapy

SUMMARY:
The goal of this controlled, randomized, clinical trial is to evaluate the effect of vinpocetine on clinical outcomes on the diabetic nephropathy patients.

The following will be evaluated; anthropometrics, kidney functions, glucose panel, lipid panel, ICAM-1, quality of life.

Participants will receive either vinpocetine or placebo, twice daily for 3 months.

DETAILED DESCRIPTION:
Diabetes mellitus affects around 537 million people globally, projected to reach over 700 million by 2045. Egypt is notably impacted, ranking tenth in prevalence and contributing significantly to chronic kidney disease, blindness, and stroke. Diabetic nephropathy (DN) arises as a severe complication, affecting about 50% of type 2 diabetes patients and leading to end-stage kidney disease. Its pathogenesis involves complex mechanisms like persistent hyperglycemia, inflammation, oxidative stress, and endothelial dysfunction, culminating in kidney damage and subsequently fibrosis.

Current treatments focus on managing blood glucose, pressure, and lipid levels, often using drugs that target the renin-angiotensin-aldosterone system. However, these therapies aren't always sufficient to prevent progression to end-stage renal disease. Therefore, exploring new approaches is crucial.

Vinpocetine, a derivative of Vinca minor leaves, is a selective inhibitor of phosphodiesterase type 1 (PDE1). It has noteworthy antioxidant, anti-inflammatory, and anti-apoptotic properties.

Clinical and experimental studies suggest its potential in various conditions, including neurodegenerative disorders, cardiovascular diseases, and inflammation-related ailments. Notably, it has shown promising effects in improving endothelial function and reducing inflammatory markers like TNF-α and IL-6.

In kidney injury models, Vinpocetine has demonstrated nephroprotective effects, improving kidney function markers, reducing albumin excretion, and decreasing renal hypertrophy. It can also exert its antioxidant effects through the restoration of the depleted GSH content, and the attenuation of the increase in MDA levels. In a clinical trial investigating the effect of vinpocetine in acute ischemic stroke patients, vinpocetine inhibited the upregulation of TNF-α, IL-6, MCP-1, ICAM-1, VCAM-1, as well as CRP in blood plasma. It also appears to impact atherosclerosis by positively affecting lipid profiles and reducing atherosclerosis lesion formation through mechanisms like inhibition of NF-κB and modulation of ox-LDL receptors.

Based on vinpocetine's promising profile and minimal reported side effects, this work aims to investigate the Vinpocetine's potential in treating diabetic nephropathy and associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Type II diabetic patients with CKD stage 3 (eGFR = 30 - 59 ml/min) or stage 4 (eGFR 15-29 ml/min),
* Albumin/Creatinine ratio (ACR): 30 - 300 μg /mg (microalbuminuria),
* Stable standard therapy for at least three months prior to inclusion in the study.

Exclusion Criteria:

* Kidney donor or recipient,
* Active malignancy,
* Pregnancy or breastfeeding,
* Known intolerance or hypersensitivity to VPN,
* Participation in other interventional trials,
* Patients with inadequate liver function (ALT and AST three times greater than the upper normal limits),
* Patients with severe comorbidities
* Patients receiving warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
level of Albuminuria | Samples will be measured at baseline and after 12 weeks
  assessment of the amount of albumin excreted in urine

SECONDARY OUTCOMES:
Albumin: creatinine ratio (ACR) | Samples will be measured at baseline and after 12 weeks
  The urine ACR is calculated by dividing the urine albumin concentration by the urine creatinine concentration to account for differences in urine volume and more closely approximate the gold standard, 24-hour urine albumin excretion.
Serum Creatinine | Samples will be measured at baseline and after 12 weeks
  assessment of the serum level of creatinine
Blood urea nitrogen | Samples will be measured at baseline and after 12 weeks
  assessment of the level of blood urea nitrogen in serum
Hemoglobin A1c | Samples will be measured at baseline and after 12 weeks
  assessment of the level of glycated hemoglobin
Fasting and postprandial blood glucose | Samples will be measured at baseline and after 12 weeks
  Evaluation of blood level glucose after 8-hrs fasting and 2-hrs postprandial
Lipid panel | Samples will be measured at baseline and after 12 weeks
  Serum Low-density Lipoprotein Cholesterol (LDL-C), High-density Lipoprotein Cholesterol (HDL-C), Total Cholesterol, Triglycerides
Body Mass index (BMI) | Samples will be measured at baseline and after 12 weeks
  The BMI will be calculated using the following formula BMI=Weight(kg)/ height(m)^2
Assessment of endothelial functions | Samples will be measured at baseline and after 12 weeks
  Serum ICAM-1 using ELISA
Quality of life (QoL) Assessment | Samples will be measured at baseline and after 12 weeks
  Quality of Life (QoL) assessment using Diabetes-39 (D-39) Questionnaire. The D-39 questionnaire is a multi-dimensional, self-administrating, diabetes-specific scale. It consists of 39 items in five domains, namely energy, and mobility (15 items), diabetes control (12 items), anxiety and worry (4 items), social and peer burden (5 items), and sexual functioning (3 items). Scores are marked on a seven-point scale ranging from 1 (not affected at all) to 7 (extremely affected).
  The raw score resulting from the summation of each dimension will then be transformed linearly to 0 to 100 scales, using the following formula:
  (Raw score - minimum value)/(maximum value - minimum value) × 100
  A score of 0 indicates the least impact on QoL, and a score of 100 indicates the maximum impact on QoL

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain Shams University Hospital, Cairo, Abbasseia
  - Ain Shams Hospitals, Cairo, Abbasseya